CLINICAL TRIAL: NCT02728505
Title: Tolerability and Safety of Two Weeks of Twice-Daily Low-Concentration Sinusurf Sinus Irrigation Solution vs. Saline Solution in Normal Subjects
Brief Title: SinuSurf vs. Saline Solution in Normal Subjects
Acronym: SinuSurf
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: NeilMed Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Rakesh Chandra, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 151479
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SinuSurf irrigation twice daily (Active Comparator): This arm is going to get low-concentration SinuSurf sinus irrigation solution, then a washout period, then standard NeilMed Sinus rinse.
  Interventions: Drug: SinuSurf irrigation twice daily; Drug: NeilMed Sinus rinse irrigation twice daily
- NeilMed Sinus rinse irrigation twice daily (Placebo Comparator): This arm is going to get standard NeilMed Sinus rinse, then a washout period, then low-concentration SinuSurf sinus irrigation solution.
  Interventions: Drug: SinuSurf irrigation twice daily; Drug: NeilMed Sinus rinse irrigation twice daily

INTERVENTIONS:
Drug: SinuSurf irrigation twice daily
Drug: NeilMed Sinus rinse irrigation twice daily

SUMMARY:
Single-center, prospective, placebo controlled trial of tolerability and safety of low-concentration SinuSurf sinus irrigation solution in normal subjects. Forty (40) healthy subjects aged 18-65 will be enrolled in the study.

DETAILED DESCRIPTION:
Rhinosinusitis, or sinusitis, is a bacterial or fungal infection in the sinuses that results from a build-up of mucus, which causes inflammation of the sinus cavities. NeilMed SinuSurf solution is a mucoactive surfactant designed to be added to NeilMed large-volume saline irrigation solution for the purpose of improving the clearance of mucus caused by sinusitis. In vitro studies have shown that topical surfactant therapies, such as SinuSurf, have been shown as an efficacious treatment of the inflammation of the sinuses (rhinosinusitis). In particular, these therapies have been shown to have antimicrobial effects, including a decrease in numbers of bacteria when used alone and an elimination of bacteria when combined with antibiotics. To date, initial safety studies of SinuSurf in an in-vitro model have confirmed a lack of toxicity to ciliary beat frequency and also a lack of toxicity in nasal explants model.

In a comparative analysis of saline and surfactant irrigation in post-operational endoscopic endonasal surgery subjects, Farag, et al. found those receiving surfactant irrigation reported more side effects and 20% of subjects on the surfactant irrigation discontinued use compared to none receiving saline. Rohrer, et al. found that surfactants, when added to saline, cleared sinus spaces significantly better than saline alone.

A previous version of SinuSurf was on the market from 2011-2012; however, it was removed from the market due to anecdotal reports of concerns regarding pain, dryness, and temporary alteration of sense of smell. While no reports of permanent alteration of sense of smell have been received, NeilMed wishes to assess the tolerability and safety of a revised, lower-concentration formulation of SinuSurf prior to re-introduction in the market. The purpose of this trial is to assess the tolerability and potential side effect profile, specifically alterations to the sense of smell, of a revised, low-concentration sinus irrigation solution in a population of normal subjects.

Healthy participants are included in this study because SinuSurf™ is an over-the-counter (OTC) product used for symptoms rather than one particular disease, just as are saline rinses. It is an over-the-counter product. One of the main outcome measures is the impact upon the sense of smell, which is already often compromised in patients with chronic nasal/sinus disease. Thus we seek to study it in patients with normal smell who also don't have other conditions that may impact sense of smell, which would potentially confound data interpretation. The dose/concentration is under patent, but involves one squirt of the "shampoo" into 240 cc of buffered nasal saline. There is anecdotal (internet) report that patients may have temporary smell loss with and that will be criteria for patient withdrawal and possibly early study termination.

The advice that SinuSurf™ not be used more than 5 days is in order to prevent patients with medical conditions that should be evaluated by physician from deferring medical advice. These warnings are typical of over the counter products. In the present study, the product will be used under the physician's oversight. The 7 days period is chosen because it is a full "week" and is conceivably a time interval over which one would expect any changes in outcome measures from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 with no sinonasal symptoms who are normosmic (as determined by UPSIT-40) and have normal anterior rhinoscopy.

Exclusion Criteria:

* Any symptom or sign of active nasal or sinus disease from UPSIT-40 or exam of ears and nose.
* UPSIT-40result that is not normosmic.
* Cystic fibrosis.
* Immunosuppression from disease or therapy (HIV, primary immune deficiency, diabetes, renal insufficiency, organ transplant, immune suppressive drug).
* History of previous Endoscopic Sinus Surgery or nasal surgery.
* Not willing to use contraception or abstain from sexual relations during trial period.
* Any woman who is currently pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Sense of smell assessed by change in UPSIT-40 score between when subjects use SinuSurf, as compared to saline control. | 5 weeks

SECONDARY OUTCOMES:
Tolerability | 5 weeks
  Patient preference as reflected in patient daily diary.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Turner, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Rakesh K. Chandra, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided